CLINICAL TRIAL: NCT04152044
Title: Elucidating the Role of Obesity, Liver Function and Pathology With Overall Outcomes in Oesophageal Cancer
Brief Title: Obesity and Liver Function in Oesophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Noel Edward Donlon, Principal Investigator, St. James's Hospital, Ireland
Other Study IDs: SJH00003
Record Dates: First submitted 2019-11-02; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Obesity; Liver Function
MeSH Terms: conditions — Obesity | interventions — Esophagectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver biopsy, Visceral and subcutaneous obesity: Those with histology and LFT's and quantificaiton of obesity
  Interventions: Other: Observation of different types of obesity and liver pathology in patients undergoing and oesophagectomy

INTERVENTIONS:
Other: Observation of different types of obesity and liver pathology in patients undergoing and oesophagectomy — Patinets undergoing surgery

SUMMARY:
There is an established link between sarcopenia and outcomes in oesophageal cancer. There is scant reports in the literature regarding the influences of different obesity in different compartments.

DETAILED DESCRIPTION:
Oesophageal cancer rates are increasing as a result of obesity in Western society. Thr investigators are evaluating the influence of viscerala dn subcutaneous obesity on overall outcomes of the participants. In addition the investigators are evaluating if there is a correlation with Liver Function Tests and liver histopathology such as steatosis on survival in participants and post operative sequele.

ELIGIBILITY:
Inclusion Criteria:

* Those undergoing oesophagectomy

Exclusion Criteria:

* patients who only had chemotherapy/chemoradiotherapy without surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: oesophageal cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 658 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 1 year
Disease free survival | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- St. James's Hospital, Dublin, IE, Ireland

IPD SHARING:
Plan to Share IPD: No